CLINICAL TRIAL: NCT04135092
Title: Single Patient Protocol: A Phase II Study Using the Administration of Autologous T-Cells Genetically Engineered to Express T-Cell Receptors Reactive Against Mutated Neoantigens in a Patient With Metastatic Cancer Plus the Administration of Pembrolizumab
Status: No longer available | Type: Expanded Access
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 209950
Record Dates: First submitted 2019-10-21; First posted 2019-10-22 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

MeSH Terms: interventions — Cyclophosphamide; fludarabine; aldesleukin; pembrolizumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Individual Patient TCR Transduced PBL — Day 0: Cells will be infused at a dose not to exceed .5e11 in 400 mL IV on the Patient Care Unit over 20-30 minutes (2-4 days after the last dose of fludarabine).
Drug: Cyclophosphamide — Days -7 and -6: Cyclophosphamide 60 mg/kg/day x 2 days IV in 250 mL D5W infused simultaneously with mesna 15 mg/kg/day over 1 hour x 2 days.
Drug: Fludarabine — Days -7 to -3: Fludarabine 25 mg/m2 /day IVPB daily over 30 minutes for 5 days.
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg IV (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 10 doses).
Drug: Pembrolizumab — Pembrolizumab 2 mg /kg IV over approximately 30 minutes on Day -2 and then every 3 weeks until time of disease progression.

SUMMARY:
Single Patient Expanded Access

DETAILED DESCRIPTION:
Background:

Please refer to National Cancer Institute Surgery Branch (NCI-SB) protocol 18-C-0049, Amendment F.

Objective:

Under Individual Patient Expanded Access, to treat a patient with metastatic prostate cancer with autologous peripheral blood lymphocytes (PBL) that have been transduced with genes encoding T-cell receptors that recognize the mutated TP53 shared oncogene in the autologous cancer.

Eligibility:

* Must have measurable, metastatic disease as assessed per RECIST v1.1 criteria.
* Must sign the informed consent document.
* Willing to sign Durable Power of Attorney Form.
* Must have all regulatory approvals prior to start of treatment.

Design:

* Please refer to NCI-SB protocol 18-C-0049, Amendment F.
* The patient will be treated with a non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine, followed by the infusion of autologous transduced PBL and then high-dose aldesleukin. The patient will also receive pembrolizumab on Day -2 prior to cell administration and additional doses every 3 weeks following cell infusion until the time of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Measurable (per RECIST v1.1 criteria), metastatic prostate cancer.
* Refractory to approved standard systemic therapy.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Willing to sign a Durable Power of Attorney Form.
* Willing to practice birth control from the time of enrollment on this study and for four months after treatment.
* Subject must be co-enrolled on protocol 03-C-0277.

Exclusion Criteria:

Not applicable.

Age Groups: Child, Adult, Older Adult